CLINICAL TRIAL: NCT02260544
Title: A Multicenter, Open Label, Balanced, Randomized, Two-treatment, Two-period, Two-sequence, Single Dose, Cross-over Bioequivalence Study of Doxorubicin Hydrochloride Liposome Injection 20mg/10mL of Dr. Reddy's Laboratories Ltd, India, With That of Doxorubicin Hydrochloride Liposome Injection 20 mg/10mL , Manufactured by: Sun Pharmaceutical Ind. Ltd, India; in Ovarian Cancer Patients Whose Disease Has Progressed or Recurred After Platinum Based Chemotherapy and Who Are Already Receiving or Scheduled to Start Therapy With the Reference Listed Drug Under Fasting Condition.
Brief Title: Bioequivalence Study of Doxorubicin Hydrochloride Liposome Injection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 591-13
Record Dates: First submitted 2014-09-22; First posted 2014-10-09 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Ovarian Epithelial Cancer Recurrent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test Product - T (Experimental): doxorubicin hydrochloride liposome ( Dr. Reddy's Lab )
  Use the test drug (doxorubicin hydrochloride liposome Injection 20mg/10mL i.e. 2mg/mL from Dr.Reddy's Laboratories Ltd., India) ; then use the reference drug ( doxorubicin hydrochloride liposome Injection 20mg/10mL i.e. 2mg/mL from Sun Pharma ) after at least 4-weeks.
  Interventions: Drug: Doxorubicin Hydrochloride Liposome Injection
- Reference Product - R (Active Comparator): doxorubicin hydrochloride liposome ( Sun Pharma )
  Use the reference drug (doxorubicin Hydrochloride Liposome Injection 20mg/10mL i.e. 2mg/mL; from Sun Pharma ) ; then use the test drug ( doxorubicin hydrochloride liposome Injection 20mg/10mL i.e. 2mg/mL from Dr.Reddy's Laboratories Ltd., India) after at least 4 weeks.
  Interventions: Drug: Doxorubicin Hydrochloride Liposome Injection

INTERVENTIONS:
Drug: Doxorubicin Hydrochloride Liposome Injection — 50mg/m2, IV on Day 1 of each cycle, On Day 1 of Cycle 2 , patients will crossover to the alternate reference or test formulation , After completion of Cycle 2 ( Day 28) , patients will be continued on the treatment of Doxorubicin Hydrochloride Liposome injection upto 4 more cycles if tolerance permits under guidance of their attending physicians.

SUMMARY:
Bioequivalence study is proposed to be carried out on patients of ovarian cancer, who are already receiving or who in the opinion of their treating physicians are candidates for Doxorubicin liposomal injection therapy .

DETAILED DESCRIPTION:
This study has sequential two stage design. Bioequivalence based on encapsulated doxorubicin will be tested at the end of stage 1. Power analysis will be performed for the primary pharmacokinetic parameters of free Doxorubicin and liposome encapsulated Doxorubicin, for all completed patients before bioequivalence evaluation. If observed power will be >= 80% then two one-sided 90% CI will be calculated for bioequivalence assessment at stage I.

If observed power will be < 80% then bioequivalence will be evaluated at stage I. If bioequivalence met then study will be stopped and if bioequivalence not met, then required additional patients will be enrolled in stage II.

Each patient will be randomized to one of the two treatment sequences ( RT or TR ) according to a randomization scheme prepared prior to the start of the trial. Serial blood samples for determination of free doxorubicin and liposomal encapsulated doxorubicin plasma concentration for PK analysis will be obtained in each cycle .

Bioequivalence Criteria : The 94.12% confidence intervals for the ratio of geometric least squares means of ln-transformed pharmacokinetic parameters Cmax, AUC0-t and AUC0-inf should be within 80.00 to125.00% to conclude the test product is bioequivalent to the reference product.

ELIGIBILITY:
Inclusion Criteria:

* Female of Indian Nationality , between 18-60n years of age
* Able to understand investigational nature of this study and give written informed consent prior to the participation in the trial.
* Patients with ovarian cancer requiring Doxorubicin and whose disease has progressed or recurred after platinum-based chemotherapy and who are already receiving or scheduled to start therapy with reference listed drug
* ECOG performance status ≤ 2
* Cardiac function ( LVEF) ≥ 50%
* patient with life expectancy of at least 3 months
* Adequate hematopoietic, renal and liver function

Exclusion Criteria:

* Prior doxorubicin exposure that would result in a total lifetime exposure of 550mg/m2 or more after four cycles of treatment .
* Pregnant or breast-feeding female
* active opportunistic infection with mycobacteria , cytomegalovirus , toxoplasma
* Impaired cardiac function including any of the following conditions within past 6 months :

  1. Unstable angina
  2. QTc prolongation or other significant ECG abnormalities
  3. Coronary artery bypass graft surgery
* History of hypersensitivity reactions attributed to a conventional formulation of doxorubicin HCl or the components of Doxorubicin Hydrochloride liposome injection.
* known brain metastasis
* HIV positive antibody or syphilis
* Patients with significantly impaired hepatic function
* Clinically significant liver and kidney disease

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2014-07; Primary Completion 2015-04 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic ( PK ) parameter : the maximum plasma doxorubicin concentration ( Cmax ) [ Time frame : 2 cycles ] | 58 days
  The study end point will use PK parameter ( Cmax ) for free doxorubicin and liposome encapsulated doxorubicin
PK parameter : the areas under the plasma concentration versus time curve calculated from 0 to the last measurable observation ( AUC 0-t) | 58 days
  The study endpoint will use the PK parameter ( AUC 0-t) for free doxorubicin and liposome encapsulated doxorubicin ( AUC 0-t)
PK parameter : the areas under the plasma concentration versus time curve extrapolated from 0 to infinity ( AUC 0-inf) | 58 days
  The study endpoint will use the PK parameter ( AUC 0-Inf) for free doxorubicin and liposome encapsulated doxorubicin

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events ( TEAEs) | 58 days

CONTACTS AND LOCATIONS:
Overall Officials: Ashis Patnaik, MBBS, MD, Study Director — Dr. Reddy's Laboratories Limited
Locations (11):
- India (11):
  - City Cancer Center, Vijaywada, Andhra Pradesh
  - Nirmal Hospital Pvt Ltd, Surat, Gujarat
  - Srinivasam Cancer Care Hospitals India Private Limited, Bangalore, Karnataka
  - Erode Cancer Center, Erode, Karnataka
  - Cancer Clinic and Nursing Home & Jasleen Hospital, Nagpur, Maharahtra
  - Curie Manavta Cancer Centre, Nashik, Maharashtra
  - Acharya HariHar Regional Cancer Centre, Cuttack, Odisha
  - Meenakshi Mission Hospital & Research Centre, Madurai, Tamil Nadu
  - Dr. G. Viswanathan Speciality Hospitals, Trichy, Tamil Nadu
  - Bibi General Hospital, Hyderabad, Telangana
  - MNJ Institute of Oncology & Regional Cancer Centre, Hyderabad, Telangana

REFERENCES:
- See also: CTRI web site India — http://ctri.nic.in/Clinicaltrials/pmaindet2.php?trialid=9255&EncHid=&userName=